CLINICAL TRIAL: NCT04519242
Title: The BFF Study- The Better to Fix or Fuse Study 'Retaining or Removing the Joint in the Foot: A Randomized Controlled Multicenter Trial of Primary Arthrodesis Versus Joint Stabilisation in Lisfranc Fracture Dislocation Midfoot Injuries
Brief Title: The BFF Study- The Better to Fix or Fuse Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL73038.096.20
Record Dates: First submitted 2020-08-13; First posted 2020-08-19 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Lisfranc Fracture; Arthrodesis; Internal Fixation; Quality of Life
MeSH Terms: conditions — Ankylosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients enrolled in the ORIF group (Active Comparator): Open reduction and internal fixation (ORIF), ORIF will be done by using bridge plate (variable angle locking plate and/or locking plate and/or dynamic compression plate - 3.5mm, 2.7mm or 2.4mm) and/or transarticular screw osteosynthesis (4.0mm cannulated screws and/or solid small fragment screws and/or HCS). For fixation, TMT4 and/or TMT5 K-wires (1.6 or 2.0mm) can be used instead.
  Interventions: Procedure: Surgery
- Patients enrolled in the PA group (Active Comparator): PA will be done by removal of the articular surface and subsequent stabilization with bridge plate (variable angle locking plate and/or locking plate and/or dynamic compression plate - 3.5mm, 2.7mm or 2.4mm) and/or transarticular screw osteosynthesis (4.0mm cannulated screws and/or solid small fragment screws and/or HCS).
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — ORIF will be done by using bridge plate (variable angle locking plate and/or locking plate and/or dynamic compression plate - 3.5mm, 2.7mm or 2.4mm) and/or transarticular screw osteosynthesis (4.0mm cannulated screws and/or solid small fragment screws and/or HCS). For fixation TMT4 and/or TMT5 K-wires (1.6 or 2.0mm) can be used instead.
  PA will be done by removal of articular surface and subsequent stabilization with bridge plate (variable angle locking plate and/or locking plate and/or dynamic compression plate - 3.5mm, 2.7mm or 2.4mm) and/or transarticular screw osteosynthesis (4.0mm cannulated screws and/or solid small fragment screws and/or HCS).
  Type and sequence of fixation of the involved rays as needed, partial or complete fixation as needed, judgement by treating surgeon.

SUMMARY:
The aim of the proposed study is to define the optimal treatment for Lisfranc fracture-dislocation, either primary arthrodesis (PA) or open reduction and internal fixation (ORIF), regarding the quality of life, complications, functional outcomes, and cost-effectiveness. The investigators hypothesize that patients will have a better quality of life and fewer complications during follow-up when undergoing a PA for unstable fracture-dislocations in the Lisfranc midfoot joints compared to ORIF. Further, the investigators expect this approach to be more cost-effective than the operative stabilization with retaining the dislocated joints, as patients will be exposed to a reduced number of reinterventions and hospital stay and/or prolonged use of pain medication.

DETAILED DESCRIPTION:
SUMMARY

Rationale: The Lisfranc injury is a complex injury of the midfoot. It can result in persistent pain and functional impairment if treated inappropriately. In Lisfranc fracture-dislocation treatment options are primary arthrodesis of the midfoot joints or open reduction and internal fixation with retaining of the midfoot joints.

Objective: The aim of the proposed study is to define optimal treatment for the Lisfranc fracture-dislocation, either primary arthrodesis or open reduction and internal fixation, in regard to the quality of life, complications, functional outcomes and cost-effectiveness. The investigators hypothesize that patients will have a better quality of life and fewer complications during follow-up when undergoing a PA for unstable fracture-dislocations in the Lisfranc midfoot joints compared to ORIF. Further, the investigators expect this approach to be more cost-effective than the operative stabilization with retaining the dislocated joints, as patients will be exposed to a reduced number of reinterventions and hospital stay and/or prolonged use of pain medication.

Study design: A multicenter prospective randomized controlled clinical trial. Study population: All patients from 18 years and older with an acute (<6 weeks) traumatic fracture-dislocation in the Lisfranc midfoot joints, displaced or unstable with weight-bearing radiographs, and are eligible for either one of the surgical procedures. In total, this study will include n=112 patients with Lisfranc fracture-dislocation.

Intervention (if applicable): Patients with Lisfranc fracture-dislocation will be randomly allocated to treatment with either PA or ORIF.

Main study parameters/endpoints: The quality of life. Secondary outcomes: complications, functional outcomes, and cost-effectiveness.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness:

The expectation of this study is that operative treatment is beneficial for the patient with an unstable Lisfranc injury. The risk of specific complications is low and generally similar in both operative treatment modalities. PA is expected to have improved results in functional scoring systems with less secondary surgical procedures compared to ORIF. Literature indicates that both treatment options from the study are accepted for Lisfranc fracture injury. No clear advantage for one treatment option is found at present in the literature.

The burden of the study seems to be not much higher compared to standard treatment because follow-up is standardized according to current trauma guidelines. The radiation exposure will not be different from the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Acute Lisfranc fracture injury (< 6 weeks after trauma)
* Displaced or unstable with weight-bearing radiographs
* Independent for activities of daily living (yes/no question)

Exclusion Criteria:

* Open Lisfranc injury
* Pure ligamentous Lisfranc injury
* Non-displaced and stable with weight-bearing radiographs
* Contra-indications for general or locoregional anesthetic techniques
* Other fractures at the ipsilateral leg
* Pre-existent abnormalities at the Lisfranc complex
* Pre-existent immobility
* Dependent on activities of daily living (due to dementia, Alzheimer, NYHA class IV angina and heart failure, oxygen-dependent COPD)
* Rheumatoid arthritis
* Pathologic fractures (metastasis, secondary osteoporosis)
* Peripheral neuropathy and/or diabetes
* Alcohol- or drug abuse preventing adequate follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
The 5 level EQ-5D version (EQ-5d-5L) questionnaire | 2-year follow up period
  This validated questionnaire (as defined by the EQ-5D-5L questionnaire) is a descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension. When the patients has no problems at the dimension, f.e. mobility, this is coded as "1".
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society Score (AOFAS) | 2 year follow up period
  The Foot and Ankle Outcome Score (FAOS) is a 42-item questionnaire of patient-relevant outcomes in five, questionnaire for patients who have musculoskeletal disorders of the upper and lower extremities, for the ankle- hindfoot, midfoot, hallux, and lesser toes.
  It incorporates both subjective and objective information. Patients report their pain, and physicians assess alignment. The patient and physician work together to complete the functional portion. Scores range from 0 to 100, with a healthy midfoot receiving 100 points.
Foot And Ankle Disability Index (FADI) | 2 year follow up period
  The Foot and Ankle Disability Index is a 34-item questionnaire divided into two subscales: the Foot and Ankle Disability Index and the Foot and Ankle Disability Index Sport. The FADI has 26 items, and the FADI Sport has 8. The FADI contains 4 pain related items and 22 activity related items. The FADI Sport contains 8 activity related items. It assesses more difficult tasks that are essential to sport.
  Each of the 34 items is scored on a 5-point Likert scale from 0 (unable to do) to 4 (no difficulty at all). The 4 pain items of the FADI are scored 0 (none) to 4 (unbearable). The FADI has a total point value of 104 points, whereas the FADI Sport has a total point value of 32 points. The FADI and FADI Sport are scored separately as percentages, with 100% representing no dysfunction.
Alignment of the foot on weight-bearing X-rays | 2 year follow up period
  Radiographs will be interpreted as follow: Instability, e.g. displacement or malalignment will be described as:
  * AP view Lateral displacement of 2nd metatarsal on intermediate cuneiform, medial margin of the second metatarsal and the middle cuneiform not aligned; TMT 1 disruption, lateral margin of the first metatarsal not aligned with the lateral margin of the medial cuneiform; Gap between 1st and 2nd metatarsal and/or ceuneiforme medialis and intermedius (>2mm);
  * 30 degree oblique view Lateral displacement of 3rd metatarsal on lateral cuneiform, lateral margin of the third metatarsal and the lateral cuneiform not aligned; Medial margin of the fourth metatarsal and cuboid not aligned;
  * lateral view Dorsal displacement of the metatarsal bases above the level of the cuneiforms.
  * any view Bony avulsion fractures between base 2nd metatarsal and cuneiforme medialis (fleck sign), and/or between cuneiforme medialis and intermedius.
Medical Consumption Questionnaire (MCQ) | 2 year follow up period
  Medical consumption is measured on the basis of 29 questions.The scoring for items starting with "How many appointments did you have ..." is as follows. The number of agreements that the respondent mentions will be adopted. When the respondent has ticked "No appointment at all" a 0 is entered. When the respondent has nothing checked, this should be considered as missing information. Data regarding care items in which a distinction is made between different types of care collected based on multiple questions. The first question about the item in question is always oneselection question. Respondents ticking "No" can skip the following questions and are referred to the next care item via the routing. The answer "No" is scoredwith a 2. The missing values for questions that can be skipped arecoded as a valid missing. Respondents who answer "Yes" are asked further to proceed with the following questions. This asks for a specification of the care item and the number of care received.
Occurrence of complications | 2 year follow up period
  most important being post-traumatic arthritis, infection, non-union
12-Item Short Form Health Survey (SF-12) | 2- year follow up period
  The SF-12 measures eight health aspects, namely physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Productivity Cost Questionnaire (PCQ) | 2-year follow up period
  Questions 1 to 3 provide information about the amount of paid work (in hours) and the number of days per week on which the person works. The latter provides insight into the average number of hours of work per working day of the respondent. This information is needed to calculate productivity loss costs.
  The questions about productivity losses form the following modules: - Absenteeism: absenteeism from paid work (questions 4 to 6) - 'Presenteeism': productivity losses during days worked (questions 7 to 9) - Productivity loss from unpaid work (questions 10 to 12).
  Absenteeism:
  The total amount of absenteeism is then calculated by multiplying the number of days absent and the number of hours per working day of the respondent.
  To calculate the costs of productivity losses, volumes are multiplied by unit cost prices.

OTHER OUTCOMES:
Amount and type of secondary procedures | 2-year follow up period
  This includes the removing of osteosynthysis materials.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Boom NAC, Stollenwerck GANL, Evers SMAA, Poeze M. Effectiveness and cost-effectiveness of primary arthrodesis versus open reduction and internal fixation in patients with Lisfranc fracture instability (The BFF Study) study protocol for a multicenter randomized controlled trial. BMC Surg. 2021 Aug 12;21(1):323. doi: 10.1186/s12893-021-01320-1. PMID 34384419